CLINICAL TRIAL: NCT02192567
Title: Phase 1, Open Label Study to Assess the Safety and Pharmacokinetics of DS-5573a in Japanese Patients With Advanced Solid Malignant Tumors
Brief Title: Open Label Study of DS-5573a
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS5573-A-J101
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Advanced Solid Malignant Tumors
Keywords: Advanced solid malignant tumor; phase 1; oncology
MeSH Terms: conditions — Neoplasms | interventions — DS-5573a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DS-5573a does escalation (step 1) and expansion (step 2) (Experimental): Step 1 of this study will follow a 3+3 study design with a starting intravenous (IV) dose of 0.1 mg/kg.
  Eight dose levels are planned, level 1: 0.1 mg/kg, level 1.5: 0.1 mg/kg, 0.3 mg/kg, level 2: 0.3 mg/kg, level 3: 1 mg/kg, level 4: 3 mg/kg, level 5: 10 mg/kg, level 6: 20 mg/kg, level 7: 30 mg/kg Step 2: 30 subjects will be enrolled and treated at the dose determined in Step 1.
  Interventions: Drug: DS-5573a

INTERVENTIONS:
Drug: DS-5573a — Step 1 of this study will use a starting intravenous (IV) dose of 0.1 mg/kg. Eight dose levels are planned, level 1: 0.1 mg/kg, level 1.5: 0.1 mg/kg, 0.3 mg/kg, level 2: 0.3 mg/kg, level 3: 1 mg/kg, level 4: 3 mg/kg, level 5: 10 mg/kg, level 6: 20 mg/kg, level 7: 30 mg/kg.
  Step 2: 30 subjects will use the dose determined in Step 1.

SUMMARY:
This is an open-label, sequential dose escalation and expansion study to evaluate the safety, and pharmacokinetics of DS-5573a in Japanese patients with advanced solid malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor that is refractory to standard treatment, or for which no standard treatment is available.
* Eastern Cooperative Oncology Group performance status(PS) of 0 or 1

Exclusion Criteria:

* Have any of the following concomitant disease or had the history of having following disease within 6 months before enrollment:

Cardiac failure (NYHA ≥ ClassIII), myocardial infarction, cerebral infarction, unstable angina, arrhythmia requiring treatment, coronary-artery/peripheral artery bypass surgery, cerebrovascular disease, pulmonary thromboembolism, uncontrolled deep-vein thrombosis or clinically severe thromboembolic event, or autoimmune disorders requiring treatment.

* Severe or uncontrolled concomitant disease.
* Clinically active brain metastases defined as symptomatic or requiring treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing dose limiting toxicities | Day 1 through Day 28
  Number of subjects experiencing dose limiting toxicities. To investigate the safety of DS-5573a reporting on frequency and seriousness of treatment emergent adverse events.
Number of subjects experiencing adverse events | Day 1 through 45 days after last dose
  Number of subjects experiencing adverse events. To investigate the safety of DS-5573a reporting on frequency and seriousness of treatment emergent adverse events.
Pharmacokinetic profile of DS-5573a | Cycle 1 - Day 1 through Cycle 8 - Day 1
  Pharmacokinetic profile of DS-5573a. [Time Frame: Cycle 1, 2, 3: Days 1, 2, 4, 8,15; Cycle 4, 5, 6, 7, 8: Day 1] To assess the pharmacokinetic profile of DS-5573a in Japanese subjects with advanced malignant solid tumors.

SECONDARY OUTCOMES:
Incidence of human anti-human antibodies (HAHA) against DS-5573a | Cycle 1 - Day 1 through Cycle 1 - Day 15.
  Incidence of human anti-human antibodies (HAHA) against DS-5573a.
Assessment of tumor response to DS-5573a using RECIST ver1.1. | week 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90
  Assessment of tumor response is conducted every 6 weeks during the study until study end or the subject discontinues participation.
Assessment of DS-5573a-related biomarkers in blood and tumor | Cycle 1 - Days 1,2 through Cycle 3 - Days 1,2
  Assessment of DS-5573a-related biomarkers in blood and tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Tamura, MD, Principal Investigator — National Cancer Center Hospital
Locations (1):
- National Cancer Center Hospital, Tokyo, Japan